CLINICAL TRIAL: NCT04621227
Title: A PHASE 1, OPEN -LABEL, FIXED SEQUENCE STUDY TO EVALUATE THE EFFECT OF TWO STEADY STATE DOSE LEVELS OF PF-06882961 ON THE PHARMACOKINETICS OF SINGLE ORAL DOSES OF ROSUVASTATIN AND MIDAZOLAM IN OTHERWISE HEALTHY ADULT PARTICIPANTS WITH OBESITY
Brief Title: Study To Evaluate The Effect Of Two Steady State Doses of PF 06882961 On Rosuvastatin And Midazolam Pharmacokinetics In Otherwise Healthy Adult Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C3421007
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity | interventions — danuglipron; Rosuvastatin Calcium; Midazolam

STUDY DESIGN:
Intervention Model Description: Crossover
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Period 1 (Other): Participants will receive the following treatments in this sequence : (i)Rosuvastatin alone (one dose of 10 mg), (ii) Midazolam alone (one dose of 2mg), (iii) PF 06882961 alone (120 mg twice daily), (iv) PF 06882961 (120 mg twice daily) + Rosuvastatin (one dose of 10mg), (v) PF 06882961 (120 mg) + Midazolam (one dose of 2 mg), (vi) PF 06882961 (200 mg) alone, (vii) PF 06882961 (200 mg) + Rosuvastatin (one dose of 10 mg), (viii) PF 06882961 (200 mg)+ Midazolam (one dose of 2 mg) in the study.
  Interventions: Drug: PF-06882961; Drug: Rosuvastatin; Drug: Midazolam

INTERVENTIONS:
Drug: PF-06882961 — 120 mg and 200 mg BID
Drug: Rosuvastatin — 10 mg single dose
Drug: Midazolam — 2mg single dose

SUMMARY:
A Phase 1 Study To Evaluate The Effect Of Two Steady State Doses of PF 06882961 On Rosuvastatin And Midazolam Pharmacokinetics In Otherwise Healthy Adult Participants With Obesity

DETAILED DESCRIPTION:
This study is designed to look at the effect of two doses of PF 06882961 (120 milligram (mg) twice a day (BID) and 200 mg BID) on the levels of one dose of rosuvastatin 10 mg and one dose of midazolam 2 mg, in otherwise healthy, adult participants with obesity. Total duration of study from screening to the telephone visit will be approximately 17 weeks, of which up to 63 days will be inpatient. All subjects take (i) Rosuvastatin alone, Midazolam alone, PF 06882961 alone (120 mg BID), PF 06882961 (120 mg BID) + Rosuvastatin, PF 06882961 (120 mg BID) + Midazolam, PF 06882961 (200 mg BID) alone, PF 06882961 (200 mg BID) + Rosuvastatin, PF 06882961 (200 mg BID)+ Midazolam in the study.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 30.0 kg/m2 and not more than 45.4 kg/m2 at Screening.
* Stable body weight, defined as <5 kg change (per participant report) for 90 days before Screening

Exclusion Criteria:

* Known prior participation in a trial involving PF-06882961.
* Known intolerance or hypersensitivity to GLP-1R agonists.
* Known hypersensitivity to rosuvastatin or midazolam.
* Diagnosis of type 1 or type 2 diabetes mellitus or secondary forms of diabetes at screening. Note: prior diagnoses of gestational diabetes during pregnancy only are eligible if they meet the other eligibility criteria
* Any lifetime history of a suicide attempt.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* Participation in a formal weight reduction program (eg, Weight Watchers) within 90 days prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421007

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants underwent Period 1 to 8 and received study interventions as follows: Period 1: rosuvastatin 10mg once daily (QD) on Day 1; Period 2: midazolam 2mg QD on Day 1; Period 3: PF-06882961 (danuglipron) 10mg twice a day (BID) on Days 1-4, 20mg BID on Days 5-8, 40mg BID on Days 9-12, 60mg BID on Days 13-16, 80mg BID on Days 17-20, 100mg BID on Days 21-24, and 120mg BID on Days 25-28; Period 4: PF-06882961 120mg BID on Days 1-4 + rosuvastatin 10mg QD on Day 1; Period 5: PF-06882961 120mg BID + midazolam 2mg QD on Day 1; Period 6: PF-06882961 140mg BID on Days 1-4, 160mg BID on Days 5-8, 180mg BID on Days 9-12, and 200mg BID on Days 13-16; Period 7: PF-06882961 200mg BID on Days 1-4 + rosuvastatin 10mg QD on Day 1; Period 8: PF-06882961 200mg BID + midazolam 2mg QD on Day 1.
Period: Period 1 (5 Days)
Arm/Group | All Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Period 2 (2 Days)
Arm/Group | All Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Period 3 (29 Days)
Arm/Group | All Participants
Started | 16
Completed | 14
Not Completed | 2
Not completed — Physician decision due to inappropriate behavior and noncompliance | 1
Not completed — Adverse Event | 1
Period: Period 4 (4 Days)
Arm/Group | All Participants
Started | 14
Completed | 14
Not Completed | 0
Period: Period 5 (1 Day)
Arm/Group | All Participants
Started | 14
Completed | 14
Not Completed | 0
Period: Period 6 (16 Days)
Arm/Group | All Participants
Started | 14
Completed | 14
Not Completed | 0
Period: Period 7 (4 Days)
Arm/Group | All Participants
Started | 14
Completed | 14
Not Completed | 0
Period: Period 8 (2 Days)
Arm/Group | All Participants
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study intervention
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.0 (11.34)
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0
  18-44 Years | 5
  45-65 Years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Black or African American | 3
  American Indian or Alaska Native | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to Last Quantifiable Concentration (AUClast) of Rosuvastatin in Periods 1, 4 and 7
Description: AUClast is area under the plasma concentration-time profile from time 0 to last quantifiable concentration.
Time Frame: At 0 (prior to rosuvastatin dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, and 72 hours post rosuvastatin dose on Day 1 in Periods 1, 4, and 7
Population: The PK parameter analysis population was defined as all participants who received at least 1 dose of rosuvastatin and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Rosuvastatin 10mg (Period 1): Participants received rosuvastatin 10mg QD on Day 1 in Period 1.
- PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4): Participants received PF-06882961 120mg BID on Days 1-4, and rosuvastatin 10mg QD on Day 1 in Period 4.
- PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7): Participants received PF-06882961 200mg BID on Days 1-4 and rosuvastatin 10mg QD on Day 1 in Period 7.
Arm/Group | Rosuvastatin 10mg (Period 1) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7)
Number analyzed (Participants) | 16 | 14 | 14
nanogram*hour per milliliter (ng*hr/mL) | 35.17 (43) | 72.15 (50) | 100.90 (40)
Statistical Analysis 1: Comparison: Rosuvastatin 10mg (Period 1) vs PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4); Comparison for AUClast (PF-06882961 120mg BID + rosuvastatin 10mg [Period 4] vs Rosuvastatin 10mg [Period 1]); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio (%) = 202.94, 90% CI 2-sided [167.14 to 246.41]
Statistical Analysis 2: Comparison: Rosuvastatin 10mg (Period 1) vs PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7); Comparison for AUClast (PF-06882961 200mg BID + rosuvastatin 10mg [Period 7] vs Rosuvastatin 10mg [Period 1]); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio (%) = 283.73, 90% CI 2-sided [233.68 to 344.51]

2. Primary Outcome: AUClast of Midazolam in Periods 2, 5 and 8
Description: AUClast is area under the plasma concentration-time profile from time 0 to last quantifiable concentration.
Time Frame: At 0 (prior to midazolam dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post midazolam dose on Day 1 in Periods 2, 5, and 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Midazolam 2mg (Period 2): Participants received midazolam 2mg QD on Day 1 in Period 2.
- PF-06882961 120mg BID + Midazolam 2mg (Period 5): Participants received PF-06882961 120mg BID and midazolam 2mg QD on Day 1 in Period 5.
- PF-06882961 200mg BID + Midazolam 2mg (Period 8): Participants received PF-06882961 200mg BID and midazolam 2mg QD on Day 1 in Period 8.
Arm/Group | Midazolam 2mg (Period 2) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) | PF-06882961 200mg BID + Midazolam 2mg (Period 8)
Number analyzed (Participants) | 16 | 14 | 13
nanogram*hour per milliliter (ng*hr/mL) | 39.24 (27) | 19.98 (49) | 20.21 (48)
Statistical Analysis 1: Comparison: Midazolam 2mg (Period 2) vs PF-06882961 120mg BID + Midazolam 2mg (Period 5); Comparison for AUClast (PF-06882961 120mg BID + midazolam 2mg [Period 5] vs Midazolam 2mg [Period 2]); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio (%) = 50.57, 90% CI 2-sided [42.27 to 60.50]
Statistical Analysis 2: Comparison: Midazolam 2mg (Period 2) vs PF-06882961 200mg BID + Midazolam 2mg (Period 8); Comparison for AUClast (PF-06882961 200mg BID + midazolam 2mg [Period 8] vs Midazolam 2mg [Period 2]); Test type: Other — The ratio and 90% confidence interval were expressed as percentages; Mixed Models Analysis; Adjusted Geometric Mean Ratio (%) = 50.56, 90% CI 2-sided [42.06 to 60.78]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; or other serious situations such as important medical events. TEAEs were events between first dose of study drug and up to follow-up visit that were absent before treatment or that worsened after treatment. AEs presented below were TEAEs. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: From first dose of study drug (Day 1) to telephone Follow Up (Days 89-96) (approximately up to 96 days)
Population: The safety analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- PF-06882961 Titration up to 120mg BID (Period 3): Participants received PF-06882961 10mg twice a day (BID) on Days 1-4, 20mg BID on Days 5-8, 40mg BID on Days 9-12, 60mg BID on Days 13-16, 80mg BID on Days 17-20, 100mg BID on Days 21-24, and 120mg BID on Days 25-28 in Period 3.
- PF-06882961 Titration up to 200mg BID (Period 6): Participants received PF-06882961 140mg BID on Days 1-4, 160mg BID on Days 5-8, 180mg BID on Days 9-12, and 200mg BID on Days 13-16 in Period 6.
Arm/Group | Rosuvastatin 10mg (Period 1) | Midazolam 2mg (Period 2) | PF-06882961 Titration up to 120mg BID (Period 3) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) | PF-06882961 Titration up to 200mg BID (Period 6) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7) | PF-06882961 200mg BID + Midazolam 2mg (Period 8)
Number analyzed (Participants) | 16 | 16 | 16 | 14 | 14 | 14 | 14 | 14
Participants
  All-causality TEAEs | 0 | 2 | 13 | 6 | 5 | 11 | 7 | 8
  Treatment-related TEAEs | 0 | 0 | 11 | 5 | 5 | 10 | 3 | 7

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline [BL] Abnormality)
Description: Safety laboratory assessments included clinical chemistry, hematology, urinalysis, and other tests. Abnormality was determined at the investigator's discretion.
Time Frame: From BL (Day 1, the last pre-dose measurement in Period 1) to Follow Up visit (Days 68-71) (approximately up to 71 days)
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable laboratory values were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Rosuvastatin 10mg (Period 1) | Midazolam 2mg (Period 2) | PF-06882961 Titration up to 120mg BID (Period 3) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) | PF-06882961 Titration up to 200mg BID (Period 6) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7) | PF-06882961 200mg BID + Midazolam 2mg (Period 8)
Number analyzed (Participants) | 16 | 16 | 16 | 14 | 14 | 14 | 14 | 14
Participants | 0 | 3 | 5 | 2 | 3 | 5 | 0 | 9

5. Secondary Outcome: Number of Participants With Vital Signs Data Meeting the Pre-defined Categorical Summarization Criteria
Description: Single, supine vital signs assessments included systolic blood pressure (BP), diastolic BP and pulse rate. Abnormality in vital signs included: pulse rate <40 beats per minute (bpm) or >120bpm; supine diastolic BP <50 millimeter of mercury (mmHg), increase and decrease in change from BL of >=20mmHg; supine systolic blood pressure <90mmHg, increase and decrease in change from BL of >=30mmHg.
Time Frame: as for outcome 4
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable vital signs data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Rosuvastatin 10mg (Period 1) | Midazolam 2mg (Period 2) | PF-06882961 Titration up to 120mg BID (Period 3) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) | PF-06882961 Titration up to 200mg BID (Period 6) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7) | PF-06882961 200mg BID + Midazolam 2mg (Period 8)
Number analyzed (Participants) | 16 | 16 | 16 | 14 | 14 | 14 | 14 | 14
Participants
  Pulse rate value <40bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate value >120bpm | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Supine diastolic BP value <50mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Supine diastolic BP change >=20mmHg increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine diastolic BP change >=20mmHg decrease | 0 | 0 | 1 | 0 | 3 | 3 | 1 | 1
  Supine systolic BP value <90mmHg | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Supine systolic BP change >=30mmHg increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine systolic BP change >=30mmHg decrease | 0 | 0 | 2 | 0 | 2 | 3 | 2 | 0

6. Secondary Outcome: Change From Baseline in Body Weight
Description: Changes from Baseline in body weight of the participants were measured.
Time Frame: At BL (Period 1 Day 1), on Period 3 Days 1, 8, 15 and 22, Period 4 Day 1, Period 6 Days 1 and 9, Period 7 Day 1, Period 8 Day 2, and at Follow Up visit (Days 68-71)
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable body weight data were analyzed.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | All Participants
Number analyzed (Participants) | 16
kilogram (kg)
  Period 3 Day 1 / PF-06882961 titration up to 120 mg BID | -1.5 (0.82)
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120 mg BID | -1.9 (1.56)
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120 mg BID | -3.3 (1.24)
  Period 3 Day 22 / PF-06882961 titration up to 120 mg BID: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120 mg BID | -4.3 (1.69)
  Period 4 Day 1 / PF-06882961 120 mg BID + rosuvastatin 10 mg: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120 mg BID + rosuvastatin 10 mg | -5.2 (1.87)
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200 mg BID | -6.1 (2.18)
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200 mg BID | -7.5 (2.49)
  Period 7 Day 1 / PF-06882961 200 mg BID + rosuvastatin 10 mg: number analyzed (Participants) | 14
  Period 7 Day 1 / PF-06882961 200 mg BID + rosuvastatin 10 mg | -9.1 (2.76)
  Period 8 Day 2 / PF-06882961 200 mg BID + midazolam 2 mg: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200 mg BID + midazolam 2 mg | -9.9 (3.15)
  Follow up: number analyzed (Participants) | 15
  Follow up | -5.7 (3.05)

7. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting the Pre-defined Categorical Summarization Criteria
Description: ECG assessments included pulse rate (PR), QT, QTcF intervals and QRS complex. ECG abnormalities criteria included: PR interval value >= 300msec, or BL >200msec and >=25% increase from BL, or BL <=200msec and >=50% increase from BL; QRS interval value >= 140msec, or percent change from BL >=50%; QTcF value >400 and <=480msec, or >480 and <=500 msec, or >500msec, or change from BL>30 and <=60msec, or change from BL >60msec.
Time Frame: as for outcome 4
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable ECG data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Rosuvastatin 10mg (Period 1) | Midazolam 2mg (Period 2) | PF-06882961 Titration up to 120mg BID (Period 3) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) | PF-06882961 Titration up to 200mg BID (Period 6) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7) | PF-06882961 200mg BID + Midazolam 2mg (Period 8)
Number analyzed (Participants) | 16 | 16 | 16 | 14 | 14 | 14 | 14 | 14
Participants
  PR interval value>=300 msec | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  PR interval %change >=25/50% (BL >200 msec and >=25% increase or BL <=200 msec and >=50% increase) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  QRS interval value>=140 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval %change >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF value >450 and <=480 msec | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0
  QTcF value >480 and <=500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF value >500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF change >30 and <=60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF change >60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Positive Response on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS was an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced any of the following 1: completed suicide, 2: suicide attempt (response of "yes" on "actual attempt"), 3: preparatory acts towards imminent suicidal behavior ("yes" on "aborted attempt", "interrupted attempt", "preparatory acts/behavior"), 4: suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts"), 7: self-injurious behavior, no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior"). In this outcome, number of participants with positive response (response of "yes") to suicidal behavior, ideation, or any self-injurious behavior were reported.
Time Frame: At BL (Period 1 Day 1), on Period 3 Days 1, 8, 15, and 22, Period 4 Day 1, Period 6 Days 1, 9, and 16, Period 8 Day 2, at Follow Up visit (Days 68-71) and Early Termination
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable C-SSRS results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 16
Participants
  BL | 0
  BL (Past 12 months) | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID (Since last visit) | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID (Since last visit): number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID (Since last visit) | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID (Since last visit): number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID (Since last visit) | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID (Since last visit): number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID (Since last visit) | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg (Since last visit): number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg (Since last visit) | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID (Since last visit): number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID (Since last visit) | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID (Since last visit): number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID (Since last visit) | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID (Since last visit): number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID (Since last visit) | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg (Since last visit): number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg (Since last visit) | 0
  Follow Up (Since last visit): number analyzed (Participants) | 15
  Follow Up (Since last visit) | 0
  Early Termination (ET) (Since last visit): number analyzed (Participants) | 1
  Early Termination (ET) (Since last visit) | 0

9. Secondary Outcome: Number of Participants With Categorical Scores on the Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is a 9 item self-report scale for the assessment of depressive symptoms. The questions included "little interest/pleasure in things", "feeling down depressed or hopeless", "trouble falling or staying asleep", "feeling tired or little energy", "poor appetite or overeating", "feeling bad about yourself", "trouble concentrating on things", "moving slowly or fidgety/restless" and "thoughts you be better off dead". Each item was scored on scale of "not at all", "several days", "more than half the days" to "nearly every day". Total score range: 0-27 (each item with scale from 0 [not at all] to 3 [nearly every day]. Higher score=greater severity).
Time Frame: as for outcome 8
Population: The analysis set included all participants assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable PHQ-9 results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 16
Participants
  BL Little Interest/Pleasure in Things: Not At All | 16
  BL Little Interest/Pleasure in Things: Several Days | 0
  BL Little Interest/Pleasure in Things: More Than Half The Days | 0
  BL Little Interest/Pleasure in Things: Nearly Every Day | 0
  BL Feeling Down Depressed or Hopeless: Not At All | 16
  BL Feeling Down Depressed or Hopeless: Several Days | 0
  BL Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  BL Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  BL Trouble Falling or Staying Asleep: Not At All | 16
  BL Trouble Falling or Staying Asleep: Several Days | 0
  BL Trouble Falling or Staying Asleep: More Than Half The Days | 0
  BL Trouble Falling or Staying Asleep: Nearly Every Day | 0
  BL Feeling Tired or Little Energy: Not At All | 16
  BL Feeling Tired or Little Energy: Several Days | 0
  BL Feeling Tired or Little Energy: More Than Half The Days | 0
  BL Feeling Tired or Little Energy: Nearly Every Day | 0
  BL Poor Appetite or Overeating: Not At All | 15
  BL Poor Appetite or Overeating: Several Days | 1
  BL Poor Appetite or Overeating: More Than Half The Days | 0
  BL Poor Appetite or Overeating: Nearly Every Day | 0
  BL Feeling Bad About Yourself: Not At All | 16
  BL Feeling Bad About Yourself: Several Days | 0
  BL Feeling Bad About Yourself: More Than Half The Days | 0
  BL Feeling Bad About Yourself: Nearly Every Day | 0
  BL Trouble Concentrating on Things: Not At All | 16
  BL Trouble Concentrating on Things: Several Days | 0
  BL Trouble Concentrating on Things: More Than Half The Days | 0
  BL Trouble Concentrating on Things: Nearly Every Day | 0
  BL Moving Slowly or Fidgety/Restless: Not At All | 16
  BL Moving Slowly or Fidgety/Restless: Several Days | 0
  BL Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  BL Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  BL Thoughts You Be Better Off Dead: Not At All | 16
  BL Thoughts You Be Better Off Dead: Several Days | 0
  BL Thoughts You Be Better Off Dead: More Than Half The Days | 0
  BL Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 1/PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Not At All | 16
  Period 3 Day 1/PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Several Days | 0
  Period 3 Day 1/PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 1/PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Not At All | 16
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Not At All | 16
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Not At All | 15
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Several Days | 1
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Not At All | 16
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Not At All | 16
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Not At All | 16
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Not At All | 16
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Not At All | 16
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 1 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Not At All | 14
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Several Days | 1
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Not At All | 14
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Several Days | 1
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: number analyzed (Participants) | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Not At All | 15
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 8 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Not At All | 14
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Several Days | 1
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Not At All | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Not At All | 14
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Several Days | 1
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Not At All | 14
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Several Days | 1
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Not At All | 13
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Several Days | 2
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Not At All | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Not At All | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Not At All | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: number analyzed (Participants) | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Not At All | 15
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 15 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Not At All | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Several Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Not At All | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Several Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Not At All | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Several Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Not At All | 13
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Several Days | 1
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Not At All | 11
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Several Days | 3
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Poor Appetite or Overeating: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Not At All | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Several Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Feeling Bad About Yourself: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Not At All | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Several Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Trouble Concentrating on Things: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Not At All | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: number analyzed (Participants) | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Not At All | 14
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Several Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 3 Day 22 / PF-06882961 titration up to 120mg BID Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Little Interest/Pleasure in Things: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Little Interest/Pleasure in Things: Not At All | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Little Interest/Pleasure in Things: Several Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Down Depressed or Hopeless: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Down Depressed or Hopeless: Not At All | 13
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Down Depressed or Hopeless: Several Days | 1
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Falling or Staying Asleep: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Falling or Staying Asleep: Not At All | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Falling or Staying Asleep: Several Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Tired or Little Energy: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Tired or Little Energy: Not At All | 11
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Tired or Little Energy: Several Days | 3
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Poor Appetite or Overeating: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Poor Appetite or Overeating: Not At All | 12
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Poor Appetite or Overeating: Several Days | 2
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Poor Appetite or Overeating: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Poor Appetite or Overeating: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Bad About Yourself: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Bad About Yourself: Not At All | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Bad About Yourself: Several Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Bad About Yourself: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Feeling Bad About Yourself: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Concentrating on Things: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Concentrating on Things: Not At All | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Concentrating on Things: Several Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Concentrating on Things: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Trouble Concentrating on Things: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Moving Slowly or Fidgety/Restless: Not At All | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Thoughts You Be Better Off Dead: number analyzed (Participants) | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Thoughts You Be Better Off Dead: Not At All | 14
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Thoughts You Be Better Off Dead: Several Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 4 Day 1 / PF-06882961 120mg BID + rosuvastatin 10mg Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Not At All | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Not At All | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Not At All | 12
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Several Days | 2
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Several Days | 1
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Not At All | 11
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Several Days | 3
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Not At All | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Not At All | 13
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Several Days | 1
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Not At All | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: number analyzed (Participants) | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Not At All | 14
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Several Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 6 Day 1 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Not At All | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Not At All | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Not At All | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Not At All | 13
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Several Days | 1
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Not At All | 12
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Several Days | 2
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Not At All | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Not At All | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Not At All | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: number analyzed (Participants) | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Not At All | 14
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Several Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 6 Day 9 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Not At All | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Several Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Not At All | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Several Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Not At All | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Several Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Not At All | 11
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Several Days | 3
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Not At All | 13
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Several Days | 1
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Poor Appetite or Overeating: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Not At All | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Several Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Feeling Bad About Yourself: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Not At All | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Several Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Trouble Concentrating on Things: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Not At All | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: number analyzed (Participants) | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Not At All | 14
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Several Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 6 Day 16 / PF-06882961 titration up to 200mg BID Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Little Interest/Pleasure in Things: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Little Interest/Pleasure in Things: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Little Interest/Pleasure in Things: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Little Interest/Pleasure in Things: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Little Interest/Pleasure in Things: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Down Depressed or Hopeless: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Down Depressed or Hopeless: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Down Depressed or Hopeless: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Falling or Staying Asleep: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Falling or Staying Asleep: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Falling or Staying Asleep: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Tired or Little Energy: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Tired or Little Energy: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Tired or Little Energy: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Tired or Little Energy: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Tired or Little Energy: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Poor Appetite or Overeating: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Poor Appetite or Overeating: Not At All | 12
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Poor Appetite or Overeating: Several Days | 1
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Poor Appetite or Overeating: More Than Half The Days | 1
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Poor Appetite or Overeating: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Bad About Yourself: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Bad About Yourself: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Bad About Yourself: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Bad About Yourself: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Feeling Bad About Yourself: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Concentrating on Things: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Concentrating on Things: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Concentrating on Things: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Concentrating on Things: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Trouble Concentrating on Things: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Moving Slowly or Fidgety/Restless: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Moving Slowly or Fidgety/Restless: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Thoughts You Be Better Off Dead: number analyzed (Participants) | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Thoughts You Be Better Off Dead: Not At All | 14
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Thoughts You Be Better Off Dead: Several Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Period 8 Day 2 / PF-06882961 200mg BID + midazolam 2mg Thoughts You Be Better Off Dead: Nearly Every Day | 0
  Follow Up Little Interest/Pleasure in Things: number analyzed (Participants) | 15
  Follow Up Little Interest/Pleasure in Things: Not At All | 15
  Follow Up Little Interest/Pleasure in Things: Several Days | 0
  Follow Up Little Interest/Pleasure in Things: More Than Half The Days | 0
  Follow Up Little Interest/Pleasure in Things: Nearly Every Day | 0
  Follow Up Feeling Down Depressed or Hopeless: number analyzed (Participants) | 15
  Follow Up Feeling Down Depressed or Hopeless: Not At All | 15
  Follow Up Feeling Down Depressed or Hopeless: Several Days | 0
  Follow Up Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  Follow Up Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  Follow Up Trouble Falling or Staying Asleep: number analyzed (Participants) | 15
  Follow Up Trouble Falling or Staying Asleep: Not At All | 15
  Follow Up Trouble Falling or Staying Asleep: Several Days | 0
  Follow Up Trouble Falling or Staying Asleep: More Than Half The Days | 0
  Follow Up Trouble Falling or Staying Asleep: Nearly Every Day | 0
  Follow Up Feeling Tired or Little Energy: number analyzed (Participants) | 15
  Follow Up Feeling Tired or Little Energy: Not At All | 15
  Follow Up Feeling Tired or Little Energy: Several Days | 0
  Follow Up Feeling Tired or Little Energy: More Than Half The Days | 0
  Follow Up Feeling Tired or Little Energy: Nearly Every Day | 0
  Follow Up Poor Appetite or Overeating: number analyzed (Participants) | 15
  Follow Up Poor Appetite or Overeating: Not At All | 15
  Follow Up Poor Appetite or Overeating: Several Days | 0
  Follow Up Poor Appetite or Overeating: More Than Half The Days | 0
  Follow Up Poor Appetite or Overeating: Nearly Every Day | 0
  Follow Up Feeling Bad About Yourself: number analyzed (Participants) | 15
  Follow Up Feeling Bad About Yourself: Not At All | 15
  Follow Up Feeling Bad About Yourself: Several Days | 0
  Follow Up Feeling Bad About Yourself: More Than Half The Days | 0
  Follow Up Feeling Bad About Yourself: Nearly Every Day | 0
  Follow Up Trouble Concentrating on Things: number analyzed (Participants) | 15
  Follow Up Trouble Concentrating on Things: Not At All | 15
  Follow Up Trouble Concentrating on Things: Several Days | 0
  Follow Up Trouble Concentrating on Things: More Than Half The Days | 0
  Follow Up Trouble Concentrating on Things: Nearly Every Day | 0
  Follow Up Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 15
  Follow Up Moving Slowly or Fidgety/Restless: Not At All | 15
  Follow Up Moving Slowly or Fidgety/Restless: Several Days | 0
  Follow Up Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  Follow Up Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  Follow Up Thoughts You Be Better Off Dead: number analyzed (Participants) | 15
  Follow Up Thoughts You Be Better Off Dead: Not At All | 15
  Follow Up Thoughts You Be Better Off Dead: Several Days | 0
  Follow Up Thoughts You Be Better Off Dead: More Than Half The Days | 0
  Follow Up Thoughts You Be Better Off Dead: Nearly Every Day | 0
  ET Little Interest/Pleasure in Things: number analyzed (Participants) | 1
  ET Little Interest/Pleasure in Things: Not At All | 1
  ET Little Interest/Pleasure in Things: Several Days | 0
  ET Little Interest/Pleasure in Things: More Than Half The Days | 0
  ET Little Interest/Pleasure in Things: Nearly Every Day | 0
  ET Feeling Down Depressed or Hopeless: number analyzed (Participants) | 1
  ET Feeling Down Depressed or Hopeless: Not At All | 1
  ET Feeling Down Depressed or Hopeless: Several Days | 0
  ET Feeling Down Depressed or Hopeless: More Than Half The Days | 0
  ET Feeling Down Depressed or Hopeless: Nearly Every Day | 0
  ET Trouble Falling or Staying Asleep: number analyzed (Participants) | 1
  ET Trouble Falling or Staying Asleep: Not At All | 1
  ET Trouble Falling or Staying Asleep: Several Days | 0
  ET Trouble Falling or Staying Asleep: More Than Half The Days | 0
  ET Trouble Falling or Staying Asleep: Nearly Every Day | 0
  ET Feeling Tired or Little Energy: number analyzed (Participants) | 1
  ET Feeling Tired or Little Energy: Not At All | 1
  ET Feeling Tired or Little Energy: Several Days | 0
  ET Feeling Tired or Little Energy: More Than Half The Days | 0
  ET Feeling Tired or Little Energy: Nearly Every Day | 0
  ET Poor Appetite or Overeating: number analyzed (Participants) | 1
  ET Poor Appetite or Overeating: Not At All | 1
  ET Poor Appetite or Overeating: Several Days | 0
  ET Poor Appetite or Overeating: More Than Half The Days | 0
  ET Poor Appetite or Overeating: Nearly Every Day | 0
  ET Feeling Bad About Yourself: number analyzed (Participants) | 1
  ET Feeling Bad About Yourself: Not At All | 1
  ET Feeling Bad About Yourself: Several Days | 0
  ET Feeling Bad About Yourself: More Than Half The Days | 0
  ET Feeling Bad About Yourself: Nearly Every Day | 0
  ET Trouble Concentrating on Things: number analyzed (Participants) | 1
  ET Trouble Concentrating on Things: Not At All | 1
  ET Trouble Concentrating on Things: Several Days | 0
  ET Trouble Concentrating on Things: More Than Half The Days | 0
  ET Trouble Concentrating on Things: Nearly Every Day | 0
  ET Moving Slowly or Fidgety/Restless: number analyzed (Participants) | 1
  ET Moving Slowly or Fidgety/Restless: Not At All | 1
  ET Moving Slowly or Fidgety/Restless: Several Days | 0
  ET Moving Slowly or Fidgety/Restless: More Than Half The Days | 0
  ET Moving Slowly or Fidgety/Restless: Nearly Every Day | 0
  ET Thoughts You Be Better Off Dead: number analyzed (Participants) | 1
  ET Thoughts You Be Better Off Dead: Not At All | 1
  ET Thoughts You Be Better Off Dead: Several Days | 0
  ET Thoughts You Be Better Off Dead: More Than Half The Days | 0
  ET Thoughts You Be Better Off Dead: Nearly Every Day | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) to telephone Follow Up (Days 89-96) (approximately up to 96 days)
Description: SAEs and non-serious AEs were recorded on the CRF. SAEs were also reported on the Clinical Trial SAE report form to Pfizer Safety within 24 hours of awareness. The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Rosuvastatin 10mg (Period 1) | Midazolam 2mg (Period 2) | PF-06882961 Titration up to 120mg BID (Period 3) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) | PF-06882961 Titration up to 200mg BID (Period 6) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7) | PF-06882961 200mg BID + Midazolam 2mg (Period 8)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/14 | 0/14 | 0/14 | 0/14 | 1/14
Other Adverse Events (participants affected / at risk) | 0/16 | 2/16 | 13/16 | 6/14 | 5/14 | 11/14 | 7/14 | 8/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10mg (Period 1) (N=16) | Midazolam 2mg (Period 2) (N=16) | PF-06882961 Titration up to 120mg BID (Period 3) (N=16) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) (N=14) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) (N=14) | PF-06882961 Titration up to 200mg BID (Period 6) (N=14) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7) (N=14) | PF-06882961 200mg BID + Midazolam 2mg (Period 8) (N=14)
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10mg (Period 1) (N=16) | Midazolam 2mg (Period 2) (N=16) | PF-06882961 Titration up to 120mg BID (Period 3) (N=16) | PF-06882961 120mg BID + Rosuvastatin 10mg (Period 4) (N=14) | PF-06882961 120mg BID + Midazolam 2mg (Period 5) (N=14) | PF-06882961 Titration up to 200mg BID (Period 6) (N=14) | PF-06882961 200mg BID + Rosuvastatin 10mg (Period 7) (N=14) | PF-06882961 200mg BID + Midazolam 2mg (Period 8) (N=14)
Nausea (Gastrointestinal disorders) | 0 | 0 | 8 | 5 | 0 | 4 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 10 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 3 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1 | 0 | 3 | 3 | 0 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 6 | 0 | 0 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT04621227/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT04621227/SAP_001.pdf